CLINICAL TRIAL: NCT04265638
Title: One-on-one Exercise Program in Adolescent and Young Adult Cancer Survivors With a Certified Clinical Cancer Exercise Specialist
Brief Title: Exercise Intervention in Adolescent and Young Adult Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, NiCole Keith, Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IUSCC-0696
Record Dates: First submitted 2019-08-05; First posted 2020-02-11 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Long-term Effects Secondary to Cancer Therapy in Adults; Pediatric Cancer
MeSH Terms: conditions — Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental)
  Interventions: Behavioral: Exercise
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Exercise — One on one exercise with a cancer exercise specialist 1 hour 3 times a week for 12 weeks.
  Arms: Exercise

SUMMARY:
Adolescent and young adult (AYA) survivors of cancer face a future of persistent medical issues across a wide spectrum of diseases One study examining health data from this cohort (ages 15-29) reported significantly higher rates of smoking, obesity, cardiovascular disease, hypertension, asthma, and poorer mental health among the cancer survivors when compared to healthy controls. Prescribed exercise has broad and far-reaching beneficial physiological effects that cut across multiple body systems and consistently improves emotional well-being, decreases fatigue and depression, and enhances quality of life. Although a growing body of evidence consistently demonstrates the physiological and psychological benefits of exercise interventions in adults with cancer, there are no studies examining the effects of individualized, prescribed, supervised exercise in pediatric, adolescent and young adult cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 15 and ≤ 39 years,
2. History of cancer
3. At least three months off of cytotoxic chemotherapy (note: hormone therapy is permitted)

Exclusion Criteria:

1. Evidence of significant liver dysfunction, congestive heart failure, cardiovascular disease
2. History of CNS tumor
3. Down's Syndrome
4. Unable to perform aerobic and/or strength exercises with full range of motion (limb immobilization, limb amputation, or surgical complications.
5. Neurological disorder
6. Baseline exercise of 30 minutes per day three times a week already being performed.

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-06-05 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Change of the Participant Evaluation of Feasibility and Acceptability Questionnaire | weeks 12 and 24
  The Participant Evaluation of Feasibility and Acceptability Questionnaire consists of 6 items arranged on a Likert scale ranging from 1- 5, and 4 additional open-ended questions designed to elicit information concerning the benefits and barriers to participating in the resistance exercise intervention.
Change of Balance Assessment | baseline, weeks 6, 12, and 24
  The BOT2 Balance subtests 5, Number 2: Walking forward on a line and Subtest 5, Number 7: Standing on One leg on a balance beam - Eyes Open will evaluate motor-control skills that are integral for maintaining posture when standing, walking, or reaching. This motor-area composite measures control and coordination of the large musculature that aids in posture and balance. Scores are assessed to determine stability dynamically and statically, on one leg and utilizing both legs, on a balance beam when the eyes are open for more than 10 seconds and if the patient can likely do so when the eyes are closed for about 5 to 10 seconds and also a twenty-four foot straight line.
Change of Cardiovascular Systems - VO2 Peak (mL·kg-1·min-1) | baseline, weeks 6, 12, and 24
  The subject's VO2 Peak (mL-kg-1-min-1) will be used to assess the cardiovascular system.
Change of Cardiovascular Systems - FEV1 | baseline, weeks 6, 12, and 24
  The subject's forced expiratory volume in one second (FEV1) will be used to assess the cardiovascular system.
  FEV1: Male = [0.0566 (ht in cm)] - [0.0233 (age)] - 4.91
Change of Cardiovascular Systems - FCV | baseline, weeks 6, 12, and 24
  The subject's estimated forced vital capacity (FVC) will be used to assess the cardiovascular system.
  FVC: Male = [0.0774 (ht in cm)] - [0.0212 (age)] - 7.75 Female = [0.0414 (ht in cm)] - [0.0232 (age)] - 2.2
Change of Fatigue | baseline, weeks 6, 12, and 24
  The Revised Piper Fatigue Scale: Fatigue will be measured using the Piper Fatigue Inventory, which evaluates total cancer-related fatigue, as well as subscales of fatigue such as affective, behavior, cognitive, mood, and sensory. There are 4 individual subscales comprise 22 items with the average score representing total fatigue. The subscales are behavioral/severity (6 items), affective meaning (5 items), sensory (5 items) and cognitive/mood (6 items). Standardized alpha for the entire scale (n = 22 items) is 0.97, indicating that some redundancy still may exist among the items. The scale ranges from 0 to 10. A score of 0 indicates that the participant shows no signs of fatigue; a score from 1 to 3 indicates mild fatigue, 4-6 indicates moderate fatigue and a score greater than 7 indicates severe fatigue.
Change of Neuropathy 15-17 year olds | baseline, weeks 6, 12, and 24
  Pediatric Total Neuropathy Score (Peds-TNS): A multidimensional instrumentused to measure peripheral neuropathy symptoms and signs in children from 15-17 years old. This instrument assesses proximal extension of numbness, tingling, and neuropathic pain, motor function, vibration and touch sensation, strength, tendon reflexes, dizziness. These parameters provide qualitative information on symptoms, nerve conduction and sensory tests on a scale of 0 for none to 4 for severe. The individual scores are added together to provide a single measure of neuropathy called a Total Neuropathy Score.
Change of Pulmonary Systems - VO2 Peak (mL·kg-1·min-1) - FEV1 | baseline, weeks 6, 12, and 24
  The subject's VO2 Peak (mL-kg-1-min-1) will be used to forced expiratory volume in one second (FEV1).
  FEV1: Male = [0.0566 (ht in cm)] - [0.0233 (age)] - 4.91
Change of Pulmonary Systems - VO2 Peak (mL·kg-1·min-1) - FVC | baseline, weeks 6, 12, and 24
  The subject's VO2 Peak (mL-kg-1-min-1) will be used to forced expiratory volume in estimated forced vital capacity (FVC).
  FVC: Male = [0.0774 (ht in cm)] - [0.0212 (age)] - 7.75 Female = [0.0414 (ht in cm)] - [0.0232 (age)] - 2.2
Change of Cancer Therapy Fatigue | baseline, weeks 6, 12, and 24
  Functional Assessment of Cancer Therapy Fatigue Scale (FACIT-F) Brief: A questionnaire assessing fatigue and anemia-related concerns in people with cancer.
Change of Neuropathy over 17 years of age | baseline, weeks 6, 12, and 24
  Total Neuropathy Score Clinical Evaluation (TNS): The best acknowledged method to assess the severity and changes in chemotherapy-induced peripheral neurotoxicity for individuals over 17. The TNSc consists of items with scores correlating significantly with the National Cancer Institute-Common Toxicity Criteria v. 2.0

SECONDARY OUTCOMES:
Depression - BDI | Baseline, weeks 12 and 24.
  Beck Depression Inventory (BDI): The BDI is a 21-item self-report rating inventory for characteristics of depression with ratings from 0 to 3, with 3 being the most intense. The BDI is for individuals 19 and older.
Depression - CDI | Baseline, weeks 12 and 24.
  Title: Children's Depression Inventory (CDI): The CDI is a 27-item scale that is self-rated and symptom-oriented. It is a validated test for children 18 and under. There are 27 items with scores ranging from 0-2, so there is a possible total score of 0-54, with 0 being no depression to 54 being the worst. The non-clinical cut off score is 19-20, which will be the one we are using.
Beck Anxiety Inventory | Baseline, weeks 12 and 24.
  The BAI is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety in children and adults. The BAI contains 21 questions, each answer being scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms. The standardized cutoffs[4] are:
  0-7: minimal anxiety 8-15: mild anxiety 16-25: moderate anxiety 26-63: severe anxiety
Measure health-related Quality of Life | Baseline, weeks 12 and 24.
  Pediatric Quality of Life Inventory (PedsQL 4.0): The PedsQL is a modular approach to measuring health-related quality of life in healthy children and adolescents and those with acute and chronic health conditions. The PedsQL integrates generic core scales and disease-specific modules into one measurement system. The 23-item PedsQL generic core scales and disease-specific scales were designed to measure the core dimensions of health as delineated by the World Health Organization, as well as role (school) functioning. This measure is tailored to 5 different age groups: however, we will only use the section designed for teens (13-18) which is made up of 23 items comprising 4 dimensions. Ferrans & Powers Quality of Life Index: Total quality of life will be measured using the Ferrans and Powers Quality of Life Index Version III and is a 66-question index designed to evaluate social, psychological, family, and health satisfaction. This assessment is valid for ages 18 and up.
Healthy Days Core Module (CDC HRQOL-4 | baseline, weeks 6, 12, and 24
  The HRQOL is a 4-question assessment of overall health, both physical and mental health. The questionnaire is scored as follows: First unhealthy days are calculated as an estimate of the overall number of days during the previous 30 days when the respondent felt that either his or her physical or mental health was not good. The score for obtaining unhealthy days is done by combining the responses to questions 2 and 3 to calculate a summary index of overall unhealthy days, with a logical maximum of 30 unhealthy days.
Pain scale | baseline, weeks 6, 12, and 24
  Visual Analogue Scale (VAS): The VAS is a validated pain measurement for individuals age seven and older. The scale is a single line with one end denoting no pain and the other, the worst pain possible. The scale was validated in 1976 with a reliability score of 0.94. The VAS is a scale of 100-mm and ratings of 0 to 4 mm can be considered no pain; 5 to 44 mm, mild pain; 45 to 74 mm, moderate pain; and 75 to 100 mm, severe pain81
Pittsburgh Sleep Quality Index Survey | baseline, weeks 6, 12, and 24
  The PSQI is a 19-item self-rated questionnaire for evaluating subjective sleep quality over the previous month. The 19 ques-tions are combined into 7 clinically-derived component scores, each weighted equally from 0-3. The 7 component scores are added to obtain a global score ranging from 0-21, with higher scores indicating worse sleep quality.
Adverse Event Pain Assessment | baseline, weeks 6, 12, and 24
  The NCI Common Terminology Criteria for Adverse Events (CTCAE) V4.02: The NCI Common Terminology Criteria for Adverse Events Version 4.02 is a descriptive scale that grades adverse events occurring after chemotherapy in cancer patients and explores the quality of life (QOL) findings among post therapy cancer patients. A grading (severity) scale is provided for each AE term. The grading scale is 0-5 with Grade 0: no signs or symptoms of the Adverse Event to Grade 5: death.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - IU Health North Hospital, Carmel, Indiana
  - Riley Hospital for Children - Indiana University, Indianapolis, Indiana
  - Indianapolis Healthplex, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Wagner C, Oeser A, Messer S, Wender A, Cryns N, Brockelmann PJ, Holtkamp U, Baumann FT, Wiskemann J, Monsef I, Scherer RW, Mishra SI, Skoetz N. Resistance training for fatigue in people with cancer. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD015518. doi: 10.1002/14651858.CD015518. PMID 39606939